CLINICAL TRIAL: NCT01491685
Title: An Observational Assessment of the Sublingual Microcirculation of Pregnant and Non-pregnant Women (Parturient Microcirculation - Phase 1)
Brief Title: Parturient Microcirculation
Status: Completed | Type: Observational
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Ronald George, Primary Investigator, MD, FRCPC, Assistant professor, IWK Health Centre
Other Study IDs: IWK1007223
Record Dates: First submitted 2011-11-01; First posted 2011-12-14 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Pregnancy; Microcirculation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Pregnant
- Non- Pregnant

SUMMARY:
This is an observational study comparing microcirculation of pregnant to non-pregnant women. "Microcirculation" means blood flow to the extremely small blood vessels in one's body. During pregnancy the amount of blood in a woman's body increases. The body responds to this increase by pumping more blood through the heart and narrowing the size of blood vessels.

There are many types of blood vessels that have different roles in the body. Larger blood vessels. Transport blood to and from body organs like the brain and liver. Small vessels (microcirculation)distributes blood to the organ tissues. The microcirculation can change blood flow and blood pressure. Microcirculation is involved in delivering oxygen and nutrients to your body, removing waste products, and regulating body temperature.

The investigators current understanding of the microcirculation in pregnant women is limited. There is a device available that can measure microcirculation. It is known as Sidestream Dark Field (SDF) imaging. It is a special type of camera that captures pictures of the microcirculation. In this study the investigators will compare the microcirculation, as seen with SDF imaging, of pregnant women to non-pregnant women. By improving the investigators understanding of maternal microcirculation the investigators are adding to the knowledge of how the pregnant body works. The investigators hope to then translate this knowledge into further studies to improve maternal and fetal outcomes through prevention and treatment of maternal low blood pressure caused by spinal anesthesia.

DETAILED DESCRIPTION:
The objectives of this observational trial are; to compare the sublingual microcirculation of pregnant subjects to that of comparable non-pregnant volunteers; to evaluate the usefulness of a non-invasive technology, SDF imaging in pregnant and non-pregnant subjects.

By improving our understanding of maternal microcirculation we not only add to the knowledge of maternal physiology, we hope to then translate this knowledge into further studies to improve maternal and fetal clinical outcomes through prevention and treatment of maternal hypotension especially in relation to spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status I-II (ASA I Healthy, ASA II - mild and controlled systemic disease)
* Pregnant: singleton, 36 - 40 weeks EGA, non-labouring
* Non- Pregnant - Healthy female volunteers who have never been pregnant, matched to pregnant patients for age ± 1 year

Exclusion Criteria:

* Obesity (BMI > 35 kg/m2)
* Hypertensive disease (Essential, gestational, or preeclampsia)
* Diabetes Mellitus Type 1
* Cardiovascular disease
* Smoker (1 cigarette or other tobacco product within 12 months)
* Caffeinated (i.e. coffee, tea, energy drink) beverage with 2 hours

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant group - women with uncomplicated, singleton, at 36 - 40 weeks gestation, non-laboring
  Non-Pregnant group - healthy nulliparous female volunteers, matched to pregnant patients for age ± 1 year
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Microvascular Flow Index (MFI) | 1 yr
  The primary outcome is the difference between the MFI of pregnant versus non-pregnant subjects.

SECONDARY OUTCOMES:
PVD | 1 yr
  Perfused vessel density
PPV | 1 yr
  Proportion of perfused vessels

CONTACTS AND LOCATIONS:
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada